## Evaluation of Wire Electrodes to Activate the Expiratory Muscles to Restore Cough / Sub-study to Spinal Cord Stimulation to Restore Cough

## IRB08-00269/IRB98-00091

NCT number: 00995215

Date of the document: August 31, 2011

Title of Document: Statistical Analysis Plan

## Sub-study to Spinal Cord Stimulation to Restore Cough

IRB sub-study#: IRB08-00269 Date Approved: 7/21/2008

Statistical Analysis Plan: The effects of spinal cord stimulation (SCS) with disc electrode and wire leads on airway pressure generation were compared. Airway pressure generation was compared for each electrode contact at each of the three spinal cord levels and in various combinations. Since monopolar SCS with the disc leads, when applied in clinical trials, resulted in airway pressure generation that approximated pressures generated with a normal maximum cough, airway pressure generation achieved during SCS with these leads served as our *gold standard* to which all comparisons were made. Data were reported as mean ± SE. Statistical analysis was performed using a repeated measures analysis of variance and paired t-test. A p value <0.05 was taken as indicative of statistical significance.